CLINICAL TRIAL: NCT04463498
Title: Sleep in Psychiatric Care: A Transdiagnostic Group-based Sleep-school as Treatment for Comorbid Insomnia
Brief Title: Sleep in Psychiatric Care (SIP): A Transdiagnostic Group-based Sleep-school as Treatment for Comorbid Insomnia
Acronym: SIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66304
Record Dates: First submitted 2020-04-06; First posted 2020-07-09 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Sleep Disorder; Insomnia Type; Psychiatric Disorders
Keywords: sleep disorders; insomnia; psychiatric disorders; bb-glasses; group-based cognitive behavioural therapy for insomnia
MeSH Terms: conditions — Sleep Wake Disorders; Mental Disorders; Sleep Initiation and Maintenance Disorders | interventions — Waiting Lists; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: All eligible participants will be informed that there may be a waitlist (length not specified) and receive a start-date without being informed that thay are in a waitlist group or not a waitlist group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- n=15, Sleep-school 8 weeks (Experimental): Patients receive treatment as usual in the psychiatric clinic combined with participation in the sleep school. They have already been given education on sleep regulation and sleep hygiene advice in the first meeting with the sleep-school facilitator.
  Interventions: Behavioral: Group-based cognitive behavioral therapy for insomnia
- n=15, Sleep-school 8 weeks and additive bb-glasses (Experimental): Patients receive treatment as usual in the psychiatric clinic combined with participation in the sleep school and additive treatment with bb-glasses. They have already been given education on sleep regulation and sleep hygiene advice in the first meeting with the sleep-school facilitator.
  Interventions: Behavioral: Group-based cognitive behavioral therapy for insomnia; Behavioral: Group-based cognitive behavioral therapy for insomnia and additive bb-glasses
- n=30 8-week wait list for sleep-school (Active Comparator): Patients receive treatment as usual in the psychiatric clinic while they wait for participation in the sleep school. They have already been given education on sleep regulation and sleep hygiene advice in the first meeting with the sleep-school facilitator.
  Interventions: Other: 8-week wait list for sleep-school

INTERVENTIONS:
Behavioral: Group-based cognitive behavioral therapy for insomnia — Sleep education, sleep restriction, stimulus control, cognitive restructuring, relaxation techniques
  Other Names: Group - CBTi
  Arms: n=15, Sleep-school 8 weeks; n=15, Sleep-school 8 weeks and additive bb-glasses
Behavioral: Group-based cognitive behavioral therapy for insomnia and additive bb-glasses — Sleep education, sleep restriction, stimulus control, cognitive restructuring, relaxation techniques, bb-glasses worn from 3 hrs before bedtime.
  Other Names: Group - CBTi & bb-glasses
  Arms: n=15, Sleep-school 8 weeks and additive bb-glasses
Other: 8-week wait list for sleep-school — Treatment as usual in a psychiatric outpatient clinic
  Other Names: Treatment as usual
  Arms: n=30 8-week wait list for sleep-school

SUMMARY:
Sleep disorders commonly co-occur with psychiatric disorders. Sleep disorders are often treated with medication or not at all in psychiatric care, although there exist a plethora of documentation of the effectiveness of sleep interventions. There is also an increase in studies showing effectiveness of sleep-interventions when the sleep disorder co-occurs with psychiatric illness. The most common and best documented treatment for insomnia is cognitive behavioral therapy for insomnia (CBTi). There is a great gap in the knowledge on how sleep disorders can be treated effectively in psychiatric care. In this project the investigators therefore seek to investigate the effect of non-pharmacological, group-based treatment in a randomized controlled trial (RCT) where sleep and psychiatric symptoms are the primary outcome measures. CBTi comprise of sleep education, sleep restriction, stimulus control and cognitive restructuring of dysfunctional thoughts about sleep.

DETAILED DESCRIPTION:
The recommended treatment for insomnia is CBTi. Recent research has proven that dark therapy, or blocking light in wavelengths <530 nm by the use of for example orange blue-blocking glasses (bb-glasses), has shown the ability to maintain melatonin production comparable to darkness and to have an additive effect in the treatment of insomnia. The investigators therefore also want to test bb-glasses as an additive treatment to CBTi for insomnia.

The sleep-school at Bjørgvin District Psychiatric Hospital (DPS) is an already established treatment since 2017. The insomnia-group gets together every other Monday from noon until 2 pm. The group is open, which means that participants start at different dates and meet people in the group that might be at the end of their CBTi treatment. Participants are patients at the general psychiatric outpatient clinic at Bjørgvin DPS. Participant have been referred to the sleep-team by their psychologist or doctor. In this RCT the investigators will carry on the same structure for the group for participants that are recruited to the RCT.

All participants have an individual consultation before joining the group where the focus is on eligibility to participate in the group-based treatment, diagnostic evaluation, receive a standardized education on sleep-regulation and sleep hygiene advice and receive a date to start the group-based CBTi treatment. In a randomized manner, they will be allocated to the sleep-school group and start the treatment on the next possible date or to a 8 week wait-list and receive a date the treatment starts. All eligible participants will be informed that there may be a waitlist and receive a start-date without being informed that thay are in a waitlist group or not a waitlist group. All participants will be treated as usual (TAU) for their psychiatric problems parallel to either sleep-school or waitlist. Participants that start sleep-school as soon as possible, are also allocated to a) ordinary group-based CBTi 8 weeks or b) group-based CBTi 8 weeks and bb-glasses. All participant will be followed up after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the sleep-school at Bjørgvin DPS psychiatric hospital
* Patients fulfilling the Diagnostic Manual for Mental Disorders (DSM-V) criteria for insomnia comorbid to moderate to severe psychiatric illness (confirmed F-diagnosis based on the International Statistical Classification of Diseases and Related Health Problems (ICD-11) diagnostic system that are used in Norway in addition to insomnia and/or scores of ≥19 on BDI and/or scores of ≥16 on BAI at the time of referral to the sleep school)

Exclusion Criteria:

* Nightwork
* Patients that do not fulfil the DSM-V criteria for insomnia comorbid to moderate to severe psychiatric illness (confirmed F-diagnosis based on the ICD-10 diagnostic system that are used in Norway in addition to insomnia and/or scores of ≥19 on BDI and/or scores of ≥16 on BAI at the time of referral to the sleep school)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia symptoms | baseline, bi-weekly and post intervention after 8 weeks, follow-up after 12 months
  Measured by the questionnaires Insomnia severity Index (ISI) and Bergen Insomnia Scale (BIS). From sleep diaries; sleep onset latency (SOL), wake after sleep onset (WASO) and sleep efficiency (SE).

SECONDARY OUTCOMES:
Changes in insomnia diagnosis | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by the Bergen Bergen Insomnia Scale (BIS). The BIS measure subjective symptoms of insomnia during the previous week and give a total score (minimum 0, maximum 42; the higher the score, the worse severity of insomnia) and a clinical incidence of insomnia diagnosis-score (yes/no)
Changes in insomnia severity | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by the Insomnia Severity Index (ISI). The ISI is a 7-item scale assessing the perceived severity of insomnia symptoms (initial, middle, terminal), the degree of satisfaction with sleep, interference with daytime functioning, noticeability of impairment, and concern caused by the sleep problems. The scale is Likert-type with 5 anchor points ranging from 0 to 4. The scale ranges from 0 to 28 and the higher the score, the more severe insomnia. The usual time frame for responding is the last 2 weeks.
Changes in Time in bed (TIB) | baseline, bi-weekly assesment and post intervention after 8 weeks, follow-up after 12 months
  Measured by sleep diary; time from bed-time to rise time
Changes in objective early morning awakening (EMA) | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Actiwatch (AW) Spectrum PLUSS. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number of average minutes early morning awakening.
Changes in objective wake after sleep onset (WASO) | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Actiwatch (AW) Spectrum PLUSS. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number of average minutes awake after sleep onset.
Changes in Early morning awakening (EMA) | baseline, bi-weekly assesment and post intervention after 8 weeks, follow-up after 12 months
  Measured by sleep diary; minutes awake before rise time
Changes in objective time in bed (TIB) | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Actiwatch (AW) Spectrum PLUSS. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number in minutes of average time in bed.
Changes in objective sleep efficiency (SE) | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Actiwatch (AW) Spectrum PLUSS. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number from 0-100% that gives average sleep efficiency.
Changes in objective total sleep length/time asleep (TST), | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Actiwatch (AW) Spectrum PLUSS. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number in minutes of average total sleep time.
Changes in Total sleep length/time asleep (TST) | baseline, bi-weekly assesment and post intervention after 8 weeks, follow-up after 12 months
  Measured by sleep diary: Time in bed minus time awake
Changes in Sleep quality (SQ) | baseline, bi-weekly assesment and post intervention after 8 weeks, follow-up after 12 months
  Measured by sleep diary; subjective assesment of sleep quality on a scale from 1=very light to 5=very deep
Changes in Daytime function (DF) | baseline, bi-weekly assesment and post intervention after 8 weeks, follow-up after 12 months
  Measured by sleep diary; subjective assesment of daytime function on a scale from 1=very good to 5=very poor
Changes in objective sleep onset latency (SOL) | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Actiwatch (AW) Spectrum PLUSS. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number of minutes of average sleep onset latency.
Changes in beliefs and attitudes about sleep | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16). The DBAS-16 measures the degree of dysfunctional beliefs about sleep with 16 items. It has 4 subscales (1) sleep-related worry and helplessness; 2) beliefs about sleep medications; 3) expectations about sleep need; and 4) beliefs about the consequences/effects of insomnia and 1 total scale score. The higher the score, the more dysfunctional beliefs about sleep.
Changes in depression | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Becks Depression Inventory -II (BDI-II). The higher the score, the more symptoms of depression
Changes in anxiety | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Becks Anxiety Inventory (BAI). The higher the score, the more symptoms of anxiety
Changes in fatigue | baseline and post intervention after 8 weeks, and at follow-up after 12 months
  Measured by Chalder fatigue Scale (CFQ). The higher the score, the more fatigued
Work status | baseline and post intervention after 8 weeks, and at follow-up after 12 months
  Status of employment/unemployment, percentage disability benefits received. Measured by Work and social adjustment scale (WSAS) and self-report.
Well-being | baseline and post intervention after 8 weeks, and at follow-up after 12 months
  Measured by World Health Organization well-being scale (WHO-5). The higher the score, the higher well-being.

OTHER OUTCOMES:
Changes in symptoms of inattention | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by the Adult attention deficit hyperactivity disorder (ADHD) Self-Rating Scale (ASRS). The scale contains the 18 symptoms of inattention, hyperactivity, and impulsivity defining ADHD according to the DSM-IV-TR and DSM-5. The severity of the symptoms are reported on a 5-point Likert-type scale (0-4 = never, rarely, sometimes, often, to very often), with a total range of 0-72. The higher the score, the more symptoms of inattention.
Changes in vigilance | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by the Conners Continuous Performance (CPT) Test 3rd Edition™ (Conners CPT 3™)
Changes in self reported emotion regulation ability | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Difficulties in Emotion Regulation Scale (DERS) which is a 18-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores suggest greater problems with emotion regulation.
Changes in degree of experienced pain | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by a visual analogue scale (VAS Pain) ranging from 0 to 10. The higher the score, the worse the pain.
Changes in symptoms of hypochondria | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by the The Whiteley Index (WI). The 14-item WI measures assess health anxiety on a likert-scale from 1="not at all" to "5=very much". The higher the score, the more severe health anxiety.
Changes in executive functions | baseline and post intervention after 8 weeks, follow-up after 12 months
  We will measure self-reported executive functions using the Behaviour Rating Inventory for Executive Functions Self-Report (BRIEF- SR)
Changes in blood pressure | baseline and post intervention after 8 weeks, follow-up after 12 months
  We will measure systolic and diastolic pressure by a digital blood pressure measurement machine.
Changes in Heart rate variability (HRV) | baseline and post intervention after 8 weeks, follow-up after 12 months
  24 -hour HRV.
Client Satisfaction | post intervention after 8 weeks
  Measured by the Client Satisfaction Questionnaire (CSQ8). The CSQ-8 is an 8-item questionnaire that measures patient satisfaction with health services, where the items are rated from 1 (very low satisfaction) to 4 (very high satisfaction). The total score ranges from 8 to 32, with higher scores indicating higher degrees of satisfaction.
Changes in sleepiness | baseline, bi-weekly assesment and post intervention after 8 weeks, follow-up after 12 months
  Measured by the Epworth Sleepiness Scale (ESS). The ESS is an 8-item scale where the respondent grades the likelihood of falling asleep or dozing off in different daily situations. The responses are graded on a 4-point likert scale 0=no likelihodd to 3=very likely. A score of 11 or higher is considered an indication of excessive daytime sleepiness.
Changes in immediate sleepiness | baseline, bi-weekly assesment and post intervention after 8 weeks, follow-up after 12 months
  Measured by the Karolinska Sleepiness Scale (KSS). The KSS measure subjective sleepiness at a specific time point (noon). The scale gives a number from 1-9 where 9 indicates "trouble staying awake" and is the worst outcome.
Suicide attempts and admittances in psychiatric wards | baseline and post intervention after 8 weeks, and at follow-up after 12 months
  Whether or not suicide has been attempted, if applicable number og attempts and whether or nor the patient has been admitted to a psychitaric ward (voluntary/forced)

CONTACTS AND LOCATIONS:
Overall Officials: Ane Wilhelmsen-Langeland, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the following individual participant data (IPD); Study protocol and Informed Consent Form (ICF)
  IPD Sharing Time Frame Definition: A description of when the IPD and any additional supporting information will become available and for how long, including the start and end dates or period of availability. This may be provided as an absolute date (for example, starting in January 2025) or as a date relative to the time when summary data are published or otherwise made available (for example, starting 6 months after publication).
  Limit: 1000 characters.
  IPD Sharing Access Criteria Definition: Describe by what access criteria IPD and any additional supporting information will be shared, including with whom, for what types of analyses, and by what mechanism. Information about who will review requests and criteria for reviewing requests may also be provided.
Supporting Information: Study Protocol, ICF
Time Frame: By August 31st 2025
Access Criteria: Not yet decided. PI will be reviewing requests.

REFERENCES:
- [Derived] Wilhelmsen-Langeland A, Saxvig IW, Gradisar M, Vagenes VA, Pallesen S, Sorensen L, Fasmer OB, Koenig J, Bjorvatn B, Osnes B. Group cognitive behavioural therapy for insomnia compared with treatment as usual for sleep problems in psychiatric care (the SIP trials): a protocol for a pragmatic, randomised controlled trial. BMJ Open. 2025 Apr 17;15(4):e090997. doi: 10.1136/bmjopen-2024-090997. PMID 40250874

DOCUMENTS (1):
  • Study Protocol (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT04463498/Prot_000.pdf